CLINICAL TRIAL: NCT01371604
Title: A Randomized, Double-Blind Study to Evaluate the Safety and Antiviral Activity of IDX184 in Combination With Pegylated Interferon and Ribavirin for 12 Weeks in Treatment-Naïve Subjects With Genotype 1 Chronic Hepatitis C Infection
Brief Title: Safety and Antiviral Activity of IDX184 in Combination With Pegylated Interferon and Ribavirin for 12 Weeks (MK-2355-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2355-005; IDX-08C-005 (Other: Idenix Protocol Number); 2011-001878-25 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; treatment-naive
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — IDX184; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDX184 50 mg + Peg-IFN/RBV (Experimental): IDX184 50 mg and matching placebo once daily plus peginterferon alfa-2a (Peg-IFN) weekly and ribavirin (RBV) daily for 12 weeks followed by Peg-IFN weekly and RBV daily for an additional 12 or 36 weeks.
  Interventions: Drug: IDX184; Biological: Peginterferon alfa-2a (Peg-IFN); Drug: Ribavirin (RBV); Drug: Placebo
- IDX184 100 mg + Peg-IFN/RBV (Experimental): IDX184 100 mg once daily plus Peg-IFN weekly and RBV daily for 12 weeks followed by Peg-IFN weekly and RBV daily for an additional 12 or 36 weeks.
  Interventions: Drug: IDX184; Biological: Peginterferon alfa-2a (Peg-IFN); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: IDX184 — IDX184 50 mg tablet administered orally
Biological: Peginterferon alfa-2a (Peg-IFN) — Peginterferon alfa-2 180 microgram prefilled syringe administered subcutaneously once weekly
  Other Names: Pegasys
Drug: Ribavirin (RBV) — Ribavirin 200 mg tablets administered orally as a divided dose twice daily. Total daily dose to administered will be 1000 or 1200 mg based on body weight.
Drug: Placebo — Matching placebo to IDX184 50 mg tablet administered orally
  Arms: IDX184 50 mg + Peg-IFN/RBV

SUMMARY:
The purpose of this study is to assess the safety and antiviral activity of IDX184 in combination with pegylated interferon and ribavirin in treatment-naïve subjects with genotype 1 chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with documented genotype 1, chronic hepatitis C infection.
* Must agree to use double-barrier method of birth control for at least 6 months after the last dose of study drugs.
* Has not received prior antiviral treatment for HCV.
* Written informed consent by participant.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Co-infected with hepatitis B virus (HBV; hepatitis B surface antigen [HBsAg] positive) and/or human immunodeficiency virus (HIV).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who experience a serious adverse event | Up to Week 16 and end of treatment (Weeks 24 or 48)
Percentage of participants who experience an adverse event | 16 weeks
Percentage of participants who experience a grade 1-4 laboratory abnormality | 16 weeks
Percentage of participants who achieve undetectable HCV ribonucleic acid (RNA) viral levels at Week 12 | Week 12

SECONDARY OUTCOMES:
Percentage of participants who achieve undetectable HCV RNA viral levels at Week 4 | Week 4
Percentage of participants who achieve undetectable HCV RNA viral levels at the end of treatment | Weeks 24 or 48
Percentage of participants who achieve sustained virologic response (SVR) | 24 weeks after the last dose (Weeks 48 or 72)
Percentage of participants who achieve HCV RNA viral levels below the lower level of quantification (LLOQ) at Week 4 | Week 4
Percentage of participants who achieve HCV RNA viral levels below LLOQ at the end of treatment | Weeks 24 or 48
Percentage of participants who achieve HCV RNA viral levels below LLOQ at follow-up (24 weeks after the last dose) | Weeks 48 or 72

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC